CLINICAL TRIAL: NCT05256134
Title: A Phase III, Multicenter, Randomized, Parallel-Group, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Gantenerumab in Participants at Risk for or at the Earliest Stages of Alzheimer's Disease
Brief Title: A Study to Evaluate the Efficacy and Safety of Gantenerumab in Participants at Risk for or at the Earliest Stages of Alzheimer's Disease (AD)
Acronym: SKYLINE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Decision to terminate development of gantenerumab for treatment of people at risk for or at earliest stages of Alzheimer disease (AD) following results of a pre-planned analysis of safety & efficacy of gantenerumab in Graduate I&II (WN29922/WN39658).
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WN42444; 2021-001184-25 (EudraCT Number)
Record Dates: First submitted 2022-01-25; First posted 2022-02-25 (Actual); Results first posted 2024-07-09 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-05

CONDITIONS: Alzheimers Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — gantenerumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Gantenerumab (Experimental): Gantenerumab will be administered as subcutaneous (SC) injection with gradual uptitration.
  Interventions: Drug: Gantenerumab
- Placebo (Placebo Comparator): Placebo will be administered as SC injection with gradual uptitration.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Gantenerumab — Gantenerumab will be administered as per the dosing schedule described in the Arm description.
  Arms: Gantenerumab
Drug: Placebo — Placebo will be administered as per the dosing schedule described in the Arm description.
  Arms: Placebo

SUMMARY:
A study to evaluate the efficacy and safety of gantenerumab in amyloid-positive, cognitively unimpaired participants at risk for or at the earliest stages of AD. The planned number of participants for this study is approximately 1200 participants randomized in a 1:1 ratio to receive either gantenerumab or placebo (600 participants randomized to gantenerumab and 600 participants randomized to placebo).

ELIGIBILITY:
Key Inclusion Criteria:

* Willing and able to comply with the study protocol and complete all aspects of the study [including cognitive and functional assessments, physical and neurological examinations, MRI, CSF collection, genotyping, and positron emission tomography (PET) imaging].
* Cognitively unimpaired with a screening clinical dementia rating global score (CDR-GS) of 0, and Repeatable Battery for the Assessment of Neuropsychological Status Delayed Memory Index (RBANS DMI) >=80.
* Evidence of cerebral amyloid accumulation.
* Participants who have an available person (referred to as a "study partner").
* Fluent in the language of the tests used at the study site.
* Adequate visual and auditory acuity, sufficient to perform neuropsychological testing (eye glasses and hearing aids are permitted).
* Agreed not to participate in other interventional research studies for the duration of this trial.
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods that result in a failure rate of <1% per year during the treatment period and for at least 17 weeks after the final dose of study treatment.

Key Exclusion Criteria:

* Any evidence of an underlying neurological or neurodegenerative condition that may lead to cognitive impairment other than AD.
* Clinical diagnosis of mild cognitive impairment (MCI), prodromal AD, or any form of dementia.
* History or presence of intracranial or intracerebral vascular malformations, aneurysm, subarachnoid hemorrhage, or intracerebral macrohemorrhage.
* History or presence of posterior reversible encephalopathy syndrome.
* History of ischemic stroke with clinical symptoms or an acute event that is consistent with a transient ischemic attack within 12 months of screening.
* History of severe, clinically significant (i.e., resulting in persistent neurologic deficit or structural brain damage) central nervous system (CNS) trauma (e.g., cerebral contusion).
* History or presence of intracranial mass lesion (e.g., glioma, meningioma) that could potentially impair cognition or lead to progressive neurological deficits.
* Infections that may affect brain function or a history of infections that resulted in neurologic sequelae [e.g., human immunodeficiency virus (HIV), syphilis, neuroborreliosis, and viral or bacterial meningitis and encephalitis].
* History of major depression, schizophrenia, schizoaffective disorder, or bipolar disorder.
* At risk for suicide.
* History of alcohol and/or substance abuse or dependence.
* History or presence of clinically significant systemic vascular disease, atrial fibrillation or heart failure.
* Within the last year, experienced unstable or clinically significant cardiovascular disease (e.g., myocardial infarction).
* Uncontrolled hypertension.
* Chronic kidney disease, indicated by creatinine clearance <30 mL/min.
* Confirmed and unexplained impaired hepatic function.
* History of, or are known to currently have an HIV infection, or hepatitis B or hepatitis C virus infection that has not been adequately treated.
* History or presence of systemic autoimmune disorders that may lead to progressive neurological impairment with associated cognitive deficits.
* Systemic immunosuppression or immunomodulation due to the continuing effects of immunosuppressant or immunomodulating medications.
* Current COVID-19 infection.
* Evidence of folic acid or vitamin B-12 deficiency.
* Any passive immunotherapy (Ig) or other long-acting biologic agent to prevent or postpone cognitive decline within 1 year of screening.
* Any other investigational treatment within 5 half-lives or 6 months (whichever is longer) prior to screening.
* Typical/Atypical anti-psychotic medications or neuroleptic medications.
* Anticoagulation medications within 3 months of screening with no plans to initiate any prior to randomization.
* Any previous treatment with cholinesterase inhibitors and N-methyl-D-aspartate receptor antagonists are exclusionary at screening.
* Pregnant or breastfeeding, or intending to become pregnant during the study or within 17 weeks after the final dose of gantenerumab.
* Impaired coagulation.
* Known history of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric, human, or humanized antibodies or fusion proteins, including gantenerumab and gantenerumab excipients.
* Participants who reside in a skilled nursing facility such as a convalescent home or long-term care facility.
* Participants who require residence in such facilities during the study may continue in the study and be followed for efficacy and safety, provided that they have a study partner who meets the study partner requirements.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-04-19 (Actual); Primary Completion 2023-03-13 (Actual); Study Completion 2023-03-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (63):
- United States (32):
  - Banner Alzheimer?s Institute, Phoenix, Arizona
  - Banner Sun Health Research Insitute, Sun City, Arizona
  - Banner Alzheimer's Institute, Tucson, Arizona
  - California Neuroscience Research Medical Group, Inc, Sherman Oaks, California
  - JEM Research LLC, Atlantis, Florida
  - Visionary Investigators Network - Neurology Aventura, Aventura, Florida
  - Bradenton Research Center, Bradenton, Florida
  - Brain Matters Research, Inc., Delray Beach, Florida
  - Neuropsychiatric Research; Center of Southwest Florida, Fort Myers, Florida
  - ClinCloud, LLC, Maitland, Florida
  - K2 Medical Research, LLC, Maitland, Florida
  - Optimus U Corp, Miami, Florida
  - Renstar Medical Research, Ocala, Florida
  - Charter Research - Winter Park/Orlando, Orlando, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Alzheimer's Research and Treatment Center, Stuart, Florida
  - Charter Research - Lady Lake/The Villages, The Villages, Florida
  - Alzheimer?s Research and Treatment Center, Wellington, Florida
  - Premiere Research Institute, West Palm Beach, Florida
  - Center for Advanced Research & Education, Gainesville, Georgia
  - Great Lakes Clinical Trials, Chicago, Illinois
  - Via Christi Research, Wichita, Kansas
  - Tandem Clinical Research, LLC, Marrero, Louisiana
  - Quest Research Institute, Farmington Hills, Michigan
  - University of Nebraska Medical Center; Dept of Neurological Sciences, Omaha, Nebraska
  - The Cognitive and Research Center of New Jersey, Springfield, New Jersey
  - Velocity Clinical Research, East Syracuse, New York
  - Alzheimer's Memory Center, Matthews, North Carolina
  - Ohio State University; College of Medicine, Columbus, Ohio
  - Senior Adults Specialty Research, Austin, Texas
  - Kerwin Medical Center, Dallas, Texas
  - Re:Cognition Health, Fairfax, Virginia
- Instituto Kremer, Córdoba, Argentina
- Australia (3):
  - KaRa Institute of Neurological Diseases, Macquarie Park, New South Wales
  - Heidelberg Repatriation Hospital; Medical and Cognitive Research Centre, Heidelberg West, Victoria
  - Australian Alzheimer's Research Foundation, Nedlands, Western Australia
- Canada (4):
  - Okanagan Clinical Trials, Kelowna, British Columbia
  - True North Clinical Research-Halifax, Halifax, Nova Scotia
  - Kawartha Centre - Redefining Healthy Aging, Peterborough, Ontario
  - Toronto Memory Program, Toronto, Ontario
- Italy (4):
  - Fondazione Santa Lucia IRCCS; Neurologia e Riabilitazione Neurologica, Rome, Lazio
  - IRCCS Ospedale San Raffaele; U.O. di Neurologia, Milan, Lombardy
  - IRCCS Neuromed; Neurologia I-Centro studio e cura delle demenze e UVA, Pozzilli, Molise
  - AO di Perugia - Ospedale S. Maria della Misericordia; Clinica Neurologica, Perugia, Umbria
- Poland (6):
  - KLIMED, Bia?ystok
  - NZOZ Vitamed, Bydgoszcz
  - NZOZ NEURO-KARD Ilkowski i Partnerzy Sp. Partn. Lek, Późna
  - Senior Sp. Z O.O. Poradnia Psychogeriatryczna, Sopot
  - Centrum Medyczne Euromedis Sp. z o.o., Szczecin
  - NZOZ WCA, Wroc?aw
- South Korea (3):
  - Dong-A University Hospital, Busan
  - Gachon University Gil Medical Center, Incheon
  - Konkuk University Medical Center, Seoul
- Spain (4):
  - Hospital Quiron de Madrid; Servicio de Neurologia, Pozuelo de Alarcón, Madrid
  - BARCELONABETA BRAIN RESEARCH CENTER (BBRC); FUNDACIÓN PASQUAL MARAGALL, Servicio de Neurologia, Barcelona
  - Fundación ACE; Servicio de Neurología, Barcelona
  - Hospital Virgen del Rocío; Servicio de Neurología, Seville
- Sweden (2):
  - Sahlgrenska Academy University,Neuroscience and Physiology;Departmt of Psychiatry and Neurochemistry, Mölndal
  - KAROLINSKA UNI HOSPITAL, HUDDINGE; Mottagning Kognitiv Forskning, M54, Stockholm
- United Kingdom (4):
  - Re-Cognition, Birmingham
  - University of Exeter; College of Medicine and Health, Exeter
  - Panthera Biopartners Sheffield, Sheffield
  - Southampton General Hospital, Southampton

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/ourmember/roche/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

REFERENCES:
- [Derived] Hibar DP, Bauer A, Rabe C, Borlinghaus N, Jethwa A, Kollmorgen G, Di Domenico A, Zetterberg H, Blennow K, Masters CL, Sperling RA, Bittner T. Elecsys pTau217 plasma immunoassay detection of amyloid pathology in clinical cohorts. Alzheimers Dement. 2026 Jan;22(1):e71009. doi: 10.1002/alz.71009. PMID 41537338
- [Derived] Bauer A, Rabe C, Schiffman C, Rose F, Respondek G, Gullotta F, Schlieker L, Jethwa A, Schrurs I, Manuilova E, Ostrowitzki S, Bittner T. Blood-based pre-screening in the SKYLINE secondary prevention Ph3 gantenerumab study. Alzheimers Dement. 2025 Oct;21(10):e70676. doi: 10.1002/alz.70676. PMID 41085131

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in this study at 12 investigative centers in Australia, Canada, and the United States from 19 April 2022 to 13 March 2023.
Pre-assignment Details: A total of 25 amyloid-positive, cognitively unimpaired participants at risk for or at the earliest stages of Alzheimer's Disease (AD) were randomized in a 1:1 ratio to receive either gantenerumab or placebo in this study.
Groups:
- Placebo: Participants received placebo subcutaneous (SC) injection for a maximum of 191 days. Participants had the option to choose between every week (Q1W) or every two weeks (Q2W) dosing regimens for the target dose. A gradual up titration was performed. Participants who chose the Q1W dosing regimen received placebo, SC every 4 weeks (Q4W) six times, and then Q2W six times, prior to reaching the target dose of Q1W. Participants who chose the Q2W dosing regimen received placebo, SC Q4W nine times, prior to reaching the target dose of Q2W. By the time the study was terminated, none of the participants had reached the target dose.
- Gantenerumab: Participants received gantenerumab SC injection for a maximum of 172 days. Participants had the option to choose between Q1W or Q2W dosing regimens for the target dose. A gradual up titration was performed. Participants who chose the Q1W dosing regimen received a dose of gantenerumab 120 milligrams (mg) SC Q4W three times, 255 mg SC Q4W three times, and 255 mg SC Q2W six times, prior to reaching the target dose of 255 mg Q1W (i.e., 1020 mg per month). Participants who chose the Q2W dosing regimen received a dose of gantenerumab 120 mg SC Q4W three times, 255 mg SC Q4W three times, and 510 mg SC Q4W three times, prior to reaching the target dose of 510 mg Q2W (i.e., 1020 mg per month). By the time the study was terminated, none of the participants had reached the target dose.
Period: Overall Study
Arm/Group | Placebo | Gantenerumab
Started | 12 | 13
Completed | 0 | 0
Not Completed | 12 | 13
Not completed — Study Terminated by Sponsor | 11 | 10
Not completed — Withdrawal by Subject | 1 | 3

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) Population included all participants randomly assigned to study treatment. Participants were grouped into the two arms (placebo or gantenerumab) according to the treatment assigned at randomization.
Groups:
- Placebo: Participants received placebo SC injection for a maximum of 191 days. Participants had the option to choose between Q1W or Q2W dosing regimens for the target dose. A gradual up titration was performed. Participants who chose the Q1W dosing regimen received placebo, SC Q4W six times, and then Q2W six times, prior to reaching the target dose of Q1W. Participants who chose the Q2W dosing regimen received placebo, SC Q4W nine times, prior to reaching the target dose of Q2W. By the time the study was terminated, none of the participants had reached the target dose.
- Gantenerumab: Participants received gantenerumab SC injection for a maximum of 172 days. Participants had the option to choose between Q1W or Q2W dosing regimens for the target dose. A gradual up titration was performed. Participants who chose the Q1W dosing regimen received a dose of gantenerumab 120 mg SC Q4W three times, 255 mg SC Q4W three times, and 255 mg SC Q2W six times, prior to reaching the target dose of 255 mg Q1W (i.e., 1020 mg per month). Participants who chose the Q2W dosing regimen received a dose of gantenerumab 120 mg SC Q4W three times, 255 mg SC Q4W three times, and 510 mg SC Q4W three times, prior to reaching the target dose of 510 mg Q2W (i.e., 1020 mg per month). By the time the study was terminated, none of the participants had reached the target dose.
- Total: Total of all reporting groups
Arm/Group | Placebo | Gantenerumab | Total
Number analyzed (Participants) | 12 | 13 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.9 (3.2) | 72.7 (4.7) | 71.8 (4.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 17
  Male | 4 | 4 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 10 | 7 | 17
  Unknown or Not Reported | 2 | 4 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 10 | 9 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 4 | 6
Baseline of Preclinical Alzheimer's Cognitive Composite-5 (PACC-5) [Mean (Standard Deviation); unit: score on a scale] — PACC-5=average of z-scores of 5 cognitive measures: Wechsler Memory Scale (WMS Logical Memory[LM] I-II)-Total Score LM II Delayed Recall; Free & Cued Selective Reminding Test -Immediate & Delayed Recall-Trials 1-3: Total Recall; Wechsler Adult Intelligence Scale-IV Coding-Total Raw Score; Mini Mental State Examination - Total Score; Category Fluency Test-3 categories-Vegetables, Fruits & Animals-Total Admissible Words. z-score=difference between assessment &mean of baseline assessments, divided by SD of baseline assessments. Z-scores range= -3to+3. Higher scores=better cognitive performance.
  score on a scale | 0.110 (0.7339) | -0.101 (0.5286) | 0.000 (0.6310)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in PACC-5 Score
Description: The PACC-5 is computed as the average of z-scores of the following cognitive measures: 1. Wechsler Memory Scale (WMS LM I-II) - Total Score LM II Delayed Recall; 2. Free & Cued Selective Reminding Test (FCSRT) -Immediate and Delayed Recall - Trials 1-3: Total Recall; 3. Wechsler Adult Intelligence Scale (WAIS) - IV Coding - Total Raw Score; 4. Mini Mental State Examination (MMSE) - Total Score; 5. Category Fluency Test (CFT) - 3 categories - Vegetables, Fruits and Animals - Total Admissible Words. The z-score was defined as the difference between the assessment and the mean of baseline assessments, divided by the standard deviation of baseline assessments. Z-scores range from -3 to +3 with higher scores indicating better cognitive performance.
Time Frame: Baseline to early termination visit (up to 225 days from start of treatment)
Population: ITT Population included all participants randomly assigned to study treatment. Participants were grouped into the two arms (placebo or gantenerumab) according to the treatment assigned at randomization. Overall number analyzed is the number of participants with data available for analyses.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Gantenerumab
Number analyzed (Participants) | 12 | 13
score on a scale | -0.052 (0.5790) | -0.119 (0.6038)

2. Secondary Outcome: Time From Randomization to Clinical Progression to Mild Cognitive Impairment (MCI) or Dementia Due to AD
Description: Time from randomization to clinical progression to mild cognitive impairment or dementia due to Alzheimer's disease was based on the diagnosis of the independent Clinical Adjudication Committee (iCAC).
Time Frame: Randomization to early termination Visit (up to 225 days from start of treatment)
Population: ITT Population included all participants randomly assigned to study treatment. Participants were grouped into the two arms (placebo or gantenerumab) according to the treatment assigned at randomization.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Placebo | Gantenerumab
Number analyzed (Participants) | 12 | 13
weeks | NA [NA to NA] — Data was not estimable as none of the participants met the diagnosis criteria for clinical progression i.e., No participant progressed to mild cognitive impairment or dementia due to Alzheimer's disease based on the diagnosis of the iCAC. | NA [NA to NA] — Data was not estimable as none of the participants met the diagnosis criteria for clinical progression i.e., No participant progressed to mild cognitive impairment or dementia due to Alzheimer's disease based on the diagnosis of the iCAC.

3. Secondary Outcome: Time to Onset of Confirmed Clinical Progression
Description: Time to onset of confirmed clinical progression was defined as the time from randomization to the first occurrence of two consecutive visits (approximately 6 months apart) with a Clinical Dementia Rating Global Score (CDR-GS) of > 0. CDR is a clinician reported (ClinRO) measure used to stage severity of AD dementia based on a semi-structured interview with participant & a reliable informant. CDR characterizes participant's level of cognitive & functional impairment across six domains (memory, orientation, judgment & problem solving, community affairs, home & hobbies, & personal care) on a 5-point rating. CDR-GS is calculated based on the Washington University CDR-assignment algorithm & characterizes a participant's level of global impairment/stage of dementia according to following categories: 0 (normal), 0.5 (very mild dementia), 1 (mild dementia), 2 (moderate dementia), & 3 (severe dementia). Score ranges from 0 to 3 & a high score on CDR-GS would indicate a high disease severity.
Time Frame: Randomization to early termination Visit (up to 225 days from start of treatment)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Placebo | Gantenerumab
Number analyzed (Participants) | 12 | 13
weeks | NA [NA to NA] — Data was not estimable as none of the participants met the criteria for confirmed clinical progression i.e., no participant had two consecutive visits (approximately 6 months apart) with a CDR-GS greater than 0. | NA [NA to NA] — Data was not estimable as none of the participants met the criteria for confirmed clinical progression i.e., no participant had two consecutive visits (approximately 6 months apart) with a CDR-GS greater than 0.

4. Secondary Outcome: Change From Baseline in the Amsterdam Instrumental Activities of Daily Living Questionnaire Short Version (A-IADL-Q-SV)
Description: A-IADL-Q-SV=observer reported (ObsRO) measure assessing participant's ability to perform instrumental activities of daily living (including household/leisure activities, use of household appliances, management of finances, etc.). A-IADL-Q-SV includes 30 items rated by study partner. Each item is divided into 2 questions=1st question asks if activity was performed by participant during past 4 weeks (Yes/No/Don't know). If performed, 2nd question captures level of difficulty while performing activity on 5-point Likert scale (no difficulty to no longer able to perform the activity). If not performed, 2nd question captures why activity was not performed (never done before, no longer able to do so due to physical problems, no longer able to do so due to difficulties with memory/planning/thinking/other, including free text response). A-IADL-Q-SV=average of all scored responses multiplied by 25. Score range=0-100. Higher scores=better functioning. Negative change from baseline=worsening.
Time Frame: Baseline to early termination visit (up to 225 days from start of treatment)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Gantenerumab
Number analyzed (Participants) | 12 | 11
score on a scale | -1.3 (3.93) | -0.4 (1.29)

5. Secondary Outcome: Change From Baseline in the Cognitive Function Instrument Acute (CFIa) Participant Version
Description: The CFIa is an outcome measure developed to assess memory-related cognitive and functional decline in non-demented elderly individuals. The CFIa is a modified version of the original CFI and differs in terms of recall period and item response options. The CFIa is computed as the sum of 14 items, rated on a 5-point Likert scale ranging from Never=0 to Always=4 and referring to the participant's current ability (most recent experience). Total scores range from 0 to 56. Higher scores indicate greater cognitive impairment. Negative change from baseline indicates improvement. The participant (PRO) and study partner (ObsRO) versions of the CFIa were used in this study.
Time Frame: Baseline to early termination visit (up to 225 days from start of treatment)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Gantenerumab
Number analyzed (Participants) | 12 | 11
score on a scale | 0.3 (4.52) | 0.9 (4.70)

6. Secondary Outcome: Change From Baseline in the CFIa Study Partner Version
Description: The CFIa is an outcome measure developed to assess memory-related cognitive and functional decline in non-demented elderly individuals. The CFIa is a modified version of the original CFI and differs in terms of recall period and item response options. The CFIa is computed as the sum of 14 items, rated on a 5-point Likert scale ranging from Never=0 to Always=4 and referring to the participant's current ability (most recent experience). Total scores range from 0 to 56. Higher scores indicate greater cognitive impairment. Negative change from baseline indicates improvement. The PRO and ObsRO versions of the CFIa were used in this study.
Time Frame: Baseline to early termination visit (up to 225 days from start of treatment)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Gantenerumab
Number analyzed (Participants) | 12 | 10
score on a scale | -0.8 (3.24) | 0.2 (5.14)

7. Secondary Outcome: Change From Baseline in the Clinical Dementia Rating Sum of Boxes (CDR-SB)
Description: The CDR is a ClinRO measure used to stage the severity of AD dementia based on a semi-structured interview with the participant and a reliable informant. The CDR characterizes the participant's level of cognitive and functional impairment across six domains (memory, orientation, judgment and problem solving, community affairs, home and hobbies, and personal care) on a 5-point rating scale in which 0 = None, 0.5 = questionable, 1 = mild, 2 = moderate, 3 = severe (with the exception of personal care, which is rated on a 4-point rating scale and excludes the questionable impairment level). The CDR-SB is calculated by summing the ratings across each of the six domains (total score: 0 to 18), with higher scores indicating greater impairment. A negative change from baseline indicates improvement.
Time Frame: Baseline to early termination visit (up to 225 days from start of treatment)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Gantenerumab
Number analyzed (Participants) | 12 | 10
score on a scale | 0.29 (0.498) | -0.05 (0.158)

8. Secondary Outcome: Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs), and Adverse Events of Special Interest (AESIs)
Description: An AE is any untoward medical occurrence in a patient or clinical study participant temporally associated with the use of a study treatment, whether or not considered related to the study treatment. A SAE is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability or incapacity, and leads to congenital anomaly or birth defect. An AESI included drug induced liver injury and suspected transmission of infectious agent via medicinal products.
Time Frame: Day 1 to safety follow-up visit (up to 310 days from start of treatment)
Population: Safety Evaluable Population included all participants randomly assigned to study treatment and who received at least 1 dose of study drug. Participants were grouped according to the treatment they received at first exposure.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Gantenerumab
Number analyzed (Participants) | 12 | 13
Participants
  AEs | 6 | 5
  SAEs | 0 | 0
  AESIs | 0 | 0

9. Secondary Outcome: Number of Participants With Anti-Drug Antibodies (ADAs) to Gantenerumab
Description: The number of ADA-positive participants after drug administration were determined for participants exposed to gantenerumab. For determining post-baseline incidence, participants were considered to be ADA-positive if they were ADA-negative or had missing data at baseline but developed an ADA response following study drug exposure, or if they were ADA-positive at baseline and the titer of 1 or more post-baseline samples was at least 4-fold higher in comparison to the titer at the baseline. As prespecified in the protocol, this outcome measure was applicable only to participants exposed to gantenerumab.
Time Frame: Day 1 to early termination visit (up to 216 days from start of treatment)
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Gantenerumab
Number analyzed (Participants) | 13
Participants | 0

10. Secondary Outcome: Number of Participants With Magnetic Resonance Imaging (MRI) Findings: Amyloid-related Imaging Abnormalities - Edema/Effusion (ARIA-E) and ARIA-Hemosiderin Deposition (ARIA-H)
Description: ARIA are an identified risk with anti-amyloid antibodies, including gantenerumab. These changes can be identified on brain MRI. In ARIA-E, (E for edema or effusion), edema can be seen in different areas of the brain on MRI, representing fluid leakage into the brain parenchyma or sulcal spaces. ARIA-H (H for hemosiderosis) are small foci of signal loss observed on MRI sequences sensitive for paramagnetic tissue properties and comprise cerebral microbleeds (small foci of bleeding in the brain parenchyma) and leptomeningeal hemosiderosis (small foci of bleeding on the surface of the brain). These changes also occur sporadically in AD.
Time Frame: Day 1 to early termination visit (up to 248 days from start of treatment)
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Gantenerumab
Number analyzed (Participants) | 12 | 13
Participants
  ARIA-E | 0 | 0
  ARIA-H | 0 | 1

11. Secondary Outcome: Number of Participants With Injection-site Reactions (ISRs)
Description: An AE is any unfavorable and unintended sign, symptom, or disease temporally associated with the use of an investigational product or other protocol-imposed intervention, regardless of attribution. Local injection reactions (or injection-site reactions) are defined as AEs related to the injection site that occur during or within 24 hours after study drug administration that are judged to be related to the study drug injection.
Time Frame: Day 1 to safety follow-up visit (up to 310 days from start of treatment)
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Gantenerumab
Number analyzed (Participants) | 12 | 13
Participants | 0 | 1

12. Secondary Outcome: Number of Participants With Post-baseline Suicidal Behaviors and Ideations as Assessed by Columbia-Suicide Severity Rating Scale (C-SSRS) Score
Description: The C-SSRS is an assessment tool used to assess the lifetime suicidality of a participant (baseline) as well as any new instances of suicidality (since last visit). The structured interview prompts recollection of suicidal ideation (SI), including the intensity of the ideation, behavior, & attempts with actual or potential lethality. Categories have binary responses (yes/no) & include: Wish to be Dead; Non-specific Active Suicidal Thoughts; Active SI with Any Methods (Not Plan) without Intent to Act; Active SI with Some Intent to Act, without Specific Plan; Active SI with Specific Plan & Intent, Preparatory Acts & Behavior; Aborted Attempt; Interrupted Attempt; Actual Attempt (non-fatal); Completed Suicide. SI or behavior is indicated by a "yes" answer to any of the listed categories. A score of 0 is assigned if no suicide risk is present. A score of 1 or higher indicates SI or behavior. Only categories with at least one participant with event are reported.
Time Frame: Day 1 to safety follow-up visit (up to 310 days from start of treatment)
Population: Safety Evaluable Population included all participants randomly assigned to study treatment and who received at least 1 dose of study drug. Participants were grouped according to the treatment they received at first exposure. Overall number analyzed is the number of participants with data available for analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Gantenerumab
Number analyzed (Participants) | 12 | 11
Participants | 1 | 0

13. Secondary Outcome: Change in Brain Amyloid Load Over Time as Measured by Amyloid Positron Emission Tomography (PET) in a Subset of Participants
Description: Brain amyloid load over time was planned to be assessed using [18F] florbetaben or [18F] flutemetamol tracers. These are PET radioligand selective to amyloid. Amyloid PET burden is measured in a composite region of interest (ROI) by using standardized uptake value ratio (SUVR) mapped to the centiloid scale. The weighted composite target region are composed of (both left and right side): frontal lobe, parietal lobe, temporal lobe lateral, cingulum posterior and anterior cingulate gyrus. The reference region used to normalize the composite region is the whole cerebellum. The centiloid scale anchor points are 0 and 100, where 0 represents a high-certainty amyloid negative scan and 100 represents the amount of global amyloid deposition found in a typical AD scan.
Time Frame: Baseline
Population: Data is not reported as no postbaseline samples were collected due to early termination of study by the sponsor.
Arm/Group | Placebo | Gantenerumab
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Change in Brain Tau Load Over Time as Measured by Tau PET in a Subset of Participants
Description: Change in tau load represents how much neurofibrillary tau pathology is present in brain assessed using PET scan. For the longitudinal tau PET assessment, [18F]-MK-6240 was used. Tau load is measured using SUVR in four composite target ROIs: Temporal composite target region included (both left & right) anterior & posterior superior temporal gyrus, posterior temporal lobe, fusiform gyrus, & middle and inferior temporal gyrus; Medial temporal composite region not including hippocampus included (both left & right): amygdala, parahippocampus & anterior medial & lateral temporal lobe; Frontal lobe (both left & right) & Parietal lobe (both left & right). Inferior cerebellar grey matter = reference region for calculating median SUVRs for all four target regions.
Time Frame: Baseline
Population: Data is not reported as no postbaseline samples were collected due to early termination of study by the sponsor.
Arm/Group | Placebo | Gantenerumab
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Change in Cerebrospinal Fluid (CSF) Amyloid (A) Peptide Beta (β): Aβ 1-42 Over Time in a Subset of Participants
Description: Amyloid beta is a peptide fragment of the amyloid precursor protein.
Time Frame: Baseline
Population: Data is not reported as no postbaseline samples were collected due to early termination of study by the sponsor.
Arm/Group | Placebo | Gantenerumab
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Change in CSF Amyloid Peptide: Aβ 1-40 Over Time in a Subset of Participants
Description: Amyloid beta is a peptide fragment of the amyloid precursor protein.
Time Frame: Baseline
Population: Data is not reported as no postbaseline samples were collected due to early termination of study by the sponsor.
Arm/Group | Placebo | Gantenerumab
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Change in CSF Neurofilament Light (NFL) Over Time in a Subset of Participants
Description: NFL is a neuronal cytoplasmic protein highly expressed in large, myelinated axons. Its levels increase in CSF proportionally to the degree of axonal damage in a variety of neurological disorders, including AD.
Time Frame: Baseline
Population: Data is not reported as no postbaseline samples were collected due to early termination of study by the sponsor.
Arm/Group | Placebo | Gantenerumab
Number analyzed (Participants) | 0 | 0

18. Secondary Outcome: Change in CSF Phosphorylated Tau (pTau) Over Time in a Subset of Participants
Description: CSF pTau is an indicator of neuronal injury and neurodegeneration. An elevation in levels specific pTau species, is thought to be a marker for progressive cellular degeneration in AD.
Time Frame: Baseline
Population: Data is not reported as no postbaseline samples were collected due to early termination of study by the sponsor.
Arm/Group | Placebo | Gantenerumab
Number analyzed (Participants) | 0 | 0

19. Secondary Outcome: Change in CSF Total Tau (tTau) Over Time in a Subset of Participants
Description: CSF biomarker tTau has been considered as a general marker of neurodegeneration. An elevation in levels of tau, is thought to be a marker for progressive cellular degeneration in AD.
Time Frame: Baseline
Population: Data is not reported as no postbaseline samples were collected due to early termination of study by the sponsor.
Arm/Group | Placebo | Gantenerumab
Number analyzed (Participants) | 0 | 0

20. Secondary Outcome: Change in Whole Brain Volume Over Time as Determined by MRI in a Subset of Participants
Description: Whole brain volume is measured by volumetric MRI (vMRI). Volumetric imaging is a three dimensional (3D) technique where all the MRI signals are collected from the entire tissue sample and imaged as a whole entity, therefore providing a high signal to noise ratio. Whole brain volume represents a summary measure of total brain parenchyma which includes the cerebrum, basal ganglia, diencephalon, and cerebellum.
Time Frame: Baseline
Population: Data is not reported as no postbaseline samples were collected due to early termination of study by the sponsor.
Arm/Group | Placebo | Gantenerumab
Number analyzed (Participants) | 0 | 0

21. Secondary Outcome: Change in Total Ventricular Volume Over Time as Determined by MRI in a Subset of Participants
Description: Total Ventricular Volume is measured by vMRI. Volumetric imaging is a 3D technique where all the MRI signals are collected from the entire tissue sample and imaged as a whole entity, therefore providing a high signal to noise ratio. Total ventricular volume represents a summary measure of total including right and left lateral ventricles, third ventricle and fourth ventricle of brain.
Time Frame: Baseline
Population: Data is not reported as no postbaseline samples were collected due to early termination of study by the sponsor.
Arm/Group | Placebo | Gantenerumab
Number analyzed (Participants) | 0 | 0

22. Secondary Outcome: Change in Hippocampal Volume Over Time as Determined by MRI in a Subset of Participants
Description: Total hippocampal volume is measured by vMRI. Volumetric imaging is a 3D technique where all the MRI signals are collected from the entire tissue sample and imaged as a whole entity, therefore providing a high signal to noise ratio. Total hippocampal volume is calculated by summing up right and left hippocampal volumes.
Time Frame: Baseline
Population: Data is not reported as no postbaseline samples were collected due to early termination of study by the sponsor.
Arm/Group | Placebo | Gantenerumab
Number analyzed (Participants) | 0 | 0

23. Other Pre Specified Outcome: Change in Blood Aβ 1-42 Over Time in All Participants
Description: Amyloid beta is a peptide fragment of the amyloid precursor protein.
Time Frame: Baseline to safety follow-up visit (up to 310 days from start of treatment)
Reporting Status: Not Posted

24. Other Pre Specified Outcome: Change in Blood Aβ 1-40 Over Time in All Participants
Description: Amyloid beta is a peptide fragment of the amyloid precursor protein.
Time Frame: Baseline to safety follow-up visit (up to 310 days from start of treatment)
Reporting Status: Not Posted

25. Other Pre Specified Outcome: Change in Blood NFL Over Time in All Participants
Description: NFL is a neuronal cytoplasmic protein highly expressed in large, myelinated axons. Its levels increase in blood proportionally to the degree of axonal damage in AD.
Time Frame: Baseline to safety follow-up visit (up to 310 days from start of treatment)
Reporting Status: Not Posted

26. Other Pre Specified Outcome: Change in Blood pTau Over Time in All Participants
Time Frame: Baseline to safety follow-up visit (up to 310 days from start of treatment)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Day 1 to safety follow-up visit (up to 310 days from start of treatment)
Description: Safety evaluable population included all participants randomly assigned to study treatment and who received at least 1 dose of study drug. Participants were grouped according to the treatment they received at first exposure.
Arm/Group | Placebo | Gantenerumab
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/13
Other Adverse Events (participants affected / at risk) | 6/12 | 5/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=12) | Gantenerumab (N=13)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thyroid disorder (Endocrine disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Injection site reaction (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0)
Vaccination site reaction (General disorders) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cardiac murmur (Investigations) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
SKYLINE study was terminated early & limited data could be collected & analyzed. Hence, no conclusions can be made on effectiveness of gantenerumab in treatment of people at risk for or at earliest stages of AD.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-02): https://cdn.clinicaltrials.gov/large-docs/34/NCT05256134/Prot_SAP_000.pdf